CLINICAL TRIAL: NCT00039286
Title: A Pilot Study To Assess The Utility Of 18F-Fluorodeoxyglucose Positron Emission Tomography (PET) In The Pre-Operative Evaluation Of Patients With Primary And Recurrent Breast Carcinoma
Brief Title: Positron Emission Tomography Before Surgery in Evaluating Women With Primary or Recurrent Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 01-134; P30CA008748 (NIH); MSKCC-01134; NCI-G02-2074
Record Dates: First submitted 2002-06-06; First posted 2003-01-27 (Estimated); Last update posted 2015-12-24 (Estimated); Status verified 2015-12

CONDITIONS: Breast Cancer
Keywords: stage II breast cancer; stage IIIA breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Magnetic Resonance Spectroscopy; Fluorodeoxyglucose F18

ARMS (1):
- Positron Emission Tomography (Experimental): Patients receive fludeoxyglucose F 18 IV. Approximately 1 hour later, patients undergo positron emission tomography imaging. Some patients may undergo a repeat scan in 4-6 months.
  Interventions: Procedure: positron emission tomography; Procedure: radionuclide imaging; Radiation: fludeoxyglucose F 18

INTERVENTIONS:
Procedure: positron emission tomography
Procedure: radionuclide imaging
Radiation: fludeoxyglucose F 18

SUMMARY:
RATIONALE: Imaging procedures such as positron emission tomography (PET) may improve the ability to detect the extent of breast cancer.

PURPOSE: Diagnostic trial to study the effectiveness of PET to detect the extent of breast cancer in women who have primary or recurrent breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the sensitivity, specificity, and accuracy of fludeoxyglucose F 18 (FDG) positron emission tomography (PET) as compared to conventional imaging in determining the extent of disease in women with primary or recurrent breast cancer.
* Determine how often clinical management and operative intervention plans for patients are altered based on these FDG-PET scan findings.
* Determine whether FDG-PET results in more accurate detection of disease in these patients.

OUTLINE: Patients receive fludeoxyglucose F 18 IV. Approximately 1 hour later, patients undergo positron emission tomography imaging. Some patients may undergo a repeat scan in 4-6 months.

PROJECTED ACCRUAL: (50 with primary disease and 50 with recurrent disease) will be accrued for this study within 1-2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of breast cancer for which surgical intervention is planned

  * Large primary breast cancer (i.e., larger than 5 cm, T3) as determined by prior biopsy, physical exam, or mammogram OR
  * Locally advanced breast cancer (T4) OR
  * Clinical suspicion of axillary nodal disease (N1-2) (i.e., stage IIB-IIIA) OR
  * Locally or regionally recurrent disease
* No locally recurrent disease that is non-invasive (i.e., ductal carcinoma in situ)
* No locally advanced disease (e.g., inflammatory breast cancer) that will be treated with neoadjuvant chemotherapy without surgery
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age:

* Not specified

Sex:

* Female

Menopausal status:

* Not specified

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

Other:

* No other malignancy except previously treated nonmelanoma skin cancer or carcinoma in situ of the cervix
* No known active infection
* No autoimmune disease or inflammatory disease (e.g., sarcoidosis or rheumatoid arthritis)
* Able to fast for 6 hours and tolerate a FDG-PET scan for the duration of the test
* Not pregnant or nursing

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* See Disease Characteristics

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* See Disease Characteristics

Max Age: 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2001-10; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Determine the sensitivity, specificity, and accuracy | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Elisa Rush Port, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States